CLINICAL TRIAL: NCT00727441
Title: A Randomized Three-arm Neoadjuvant and Adjuvant Feasibility and Toxicity Study of a GM-CSF Secreting Allogeneic Pancreatic Cancer Vaccine Administered Either Alone or in Combination With Either a Single Intravenous Dose or Daily Metronomic Oral Doses of Cyclophosphamide for the Treatment of Patients With Surgically Resected Adenocarcinoma of the Pancreas
Brief Title: Vaccine Therapy With or Without Cyclophosphamide in Treating Patients Undergoing Chemotherapy and Radiation Therapy for Stage I or Stage II Pancreatic Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0810; P30CA006973 (NIH); J0810; CDR0000600355; NA_00015858 (Other: JHM IRB)
Record Dates: First submitted 2008-08-01; First posted 2008-08-04 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Patients receive GVAX pancreatic cancer vaccine intradermally (ID) on day 1 of Cycle 1 and undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive an additional dose of the vaccine (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1. Treatment with the vaccine repeats every 28 days for 4 additional cycles.
  Interventions: Biological: GVAX pancreatic cancer vaccine
- Arm B (Experimental): Patients receive low-dose cyclophosphamide IV on day 0 and GVAX pancreatic cancer vaccine ID on day 1 of Cycle 1. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine on day 1. Treatment with cyclophosphamide and the vaccine repeats every 28 days for 4 additional cycles..
  Interventions: Biological: GVAX pancreatic cancer vaccine; Drug: cyclophosphamide
- Arm C (Experimental): Patients receive GVAX pancreatic cancer vaccine ID on day 1 of Cycle 1 and low-dose oral cyclophosphamide twice daily on days 1-7. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21 (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21. Treatment with the vaccine and cyclophosphamide repeats every 28 days for 4 additional cycles.
  Interventions: Biological: GVAX pancreatic cancer vaccine; Drug: cyclophosphamide

INTERVENTIONS:
Biological: GVAX pancreatic cancer vaccine — Given intradermally
Drug: cyclophosphamide — Given IV (Arm B), given orally (Arm C)
  Arms: Arm B; Arm C

SUMMARY:
RATIONALE: Vaccines made from gene-modified tumor cells may help the body build an effective immune response to kill pancreatic cancer cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vaccine therapy together with cyclophosphamide may kill more tumor cells. It is not yet known whether vaccine therapy is more effective with or without cyclophosphamide in treating patients with pancreatic cancer.

PURPOSE: This randomized clinical trial is studying the side effects of vaccine therapy and to see how well it works when given with or without cyclophosphamide in treating patients undergoing chemotherapy and radiation therapy for stage I or stage II pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and feasibility of a GVAX pancreatic cancer vaccine (GM-CSF gene-transfected allogeneic pancreatic cancer vaccine) when administered alone or in combination with a single intravenous dose or daily metronomic oral doses of cyclophosphamide as neoadjuvant and adjuvant treatment in patients with resectable stage I or II adenocarcinoma of the head, neck, or uncinate process of the pancreas.
* To assess the immune cell infiltrates, particularly T-regulatory cells (Tregs) and CD4+ and CD8+ effector T cells, after neoadjuvant GVAX pancreatic cancer vaccination.
* To assess the changes in the number and function of peripheral mesothelin-specific CD8+ T cells and CD4+, FoxP3+, and GITR+ Tregs after each GVAX pancreatic cancer vaccination when administered alone or in combination with a single dose or metronomic doses of cyclophosphamide.

Secondary

* To estimate disease-free and overall survival of patients treated with these regimens.
* To estimate the effect of immune parameters on disease-free and overall survival of these patients.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

* Arm A: Patients receive GVAX pancreatic cancer vaccine intradermally (ID) on day 1 and undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive an additional dose of the vaccine. Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1. Treatment with the vaccine repeats every 28 days for 4 courses.
* Arm B: Patients receive low-dose cyclophosphamide IV on day 0 and GVAX pancreatic cancer vaccine ID on day 1. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine on day 1. Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine on day 1. Treatment with cyclophosphamide and the vaccine repeats every 28 days for 4 courses.
* Arm C: Patients receive GVAX pancreatic cancer vaccine ID on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21. Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21. Treatment with the vaccine and cyclophosphamide repeats every 28 days for 4 courses.

Patients undergo blood sample collection periodically for correlative laboratory studies, including immune cell analysis. Immune cell analysis includes monitoring the quantitative change of peripheral blood lymphocytes, including regulatory T cells (Tregs), and functional analysis of T-cell immune response. Tumor tissue samples collected at the time of surgery are analyzed for tumor antigens and infiltrating immune cells by immunohistochemistry and quantitative real-time PCR.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed adenocarcinoma of the head, neck, or uncinate process of the pancreas

  * Stage I or II disease
* Surgically resectable disease (R0 or R1) by spiral CT scan

  * No distant metastases
  * A clear fat plane is present around the celiac and superior mesenteric arteries
  * Patent superior mesenteric and portal veins
* Candidate for a pancreaticoduodenectomy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Hemoglobin ≥ 9 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 2 mg/dL
* AST and ALT ≤ 2 times upper limit of normal (ULN)
* Amylase ≤ 2 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Hyperbilirubinemia secondary to tumor-associated extrahepatic biliary obstruction allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 4 weeks after the completion of study treatment
* No history of autoimmune disease, including systemic lupus erythematosus, sarcoidosis, rheumatoid arthritis, glomerulonephritis, or vasculitis
* No uncontrolled medical problems
* No active infections
* No other cancer within the past 5 years except for superficial bladder cancer, nonmelanoma skin cancer, or low-grade prostate cancer not requiring therapy

PRIOR CONCURRENT THERAPY:

* More than 28 days since prior anticancer therapy
* No prior cancer immunotherapy, including the same pancreatic cancer vaccine used in this study
* More than 28 days since prior systemic steroid therapy or immunosuppressive therapy
* No systemic steroid therapy or immunosuppressive therapy during and within 28 days after vaccine administration
* No other concurrent immunotherapy, chemotherapy, radiotherapy, gene therapy, biologic therapy, or investigational therapy for the treatment of pancreatic cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-07-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Laheru, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - GVAX Vaccine Without Cyclophosphamide: Patients receive GVAX pancreatic cancer vaccine intradermally (ID) on day 1 of Cycle 1 and undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive an additional dose of the vaccine (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1. Treatment with the vaccine repeats every 28 days for 4 additional cycles.
  GVAX pancreatic cancer vaccine: Given intradermally
- Arm B - GVAX Vaccine With IV Cyclophosphamide: Patients receive low-dose cyclophosphamide IV on day 0 and GVAX pancreatic cancer vaccine ID on day 1 of Cycle 1. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine on day 1. Treatment with cyclophosphamide and the vaccine repeats every 28 days for 4 additional cycles..
  GVAX pancreatic cancer vaccine: Given intradermally
  Cyclophosphamide: Given IV
- Arm C - GVAX Vaccine With PO Cyclophosphamide: Patients receive GVAX pancreatic cancer vaccine ID on day 1 of Cycle 1 and low-dose oral cyclophosphamide twice daily on days 1-7. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21 (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21. Treatment with the vaccine and cyclophosphamide repeats every 28 days for 4 additional cycles.
  GVAX pancreatic cancer vaccine: Given intradermally
  Cyclophosphamide: Given orally
Period: Overall Study
Arm/Group | Arm A - GVAX Vaccine Without Cyclophosphamide | Arm B - GVAX Vaccine With IV Cyclophosphamide | Arm C - GVAX Vaccine With PO Cyclophosphamide
Started | 29 | 28 | 30
Completed | 11 | 6 | 5
Not Completed | 18 | 22 | 25
Not completed — Disease Progression | 11 | 14 | 17
Not completed — Eligibility | 7 | 5 | 7
Not completed — Death | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B - GVAX Vaccine With IV Cyclophosphamide: Patients receive low-dose cyclophosphamide IV on day 0 and GVAX pancreatic cancer vaccine ID on day 1 of Cycle 1. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive low-dose cyclophosphamide IV on day 0 and the vaccine on day 1. Treatment with cyclophosphamide and the vaccine repeats every 28 days for 4 additional cycles..
  GVAX pancreatic cancer vaccine: Given intradermally
  cyclophosphamide: Given IV (Arm B), given orally (Arm C)
- Arm C - GVAX Vaccine With PO Cyclophosphamide: Patients receive GVAX pancreatic cancer vaccine ID on day 1 of Cycle 1 and low-dose oral (PO) cyclophosphamide twice daily on days 1-7. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21 (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21. Treatment with the vaccine and cyclophosphamide repeats every 28 days for 4 additional cycles.
  GVAX pancreatic cancer vaccine: Given intradermally
  cyclophosphamide: Given IV (Arm B), given orally (Arm C)
- Total: Total of all reporting groups
Arm/Group | Arm A - GVAX Vaccine Without Cyclophosphamide | Arm B - GVAX Vaccine With IV Cyclophosphamide | Arm C - GVAX Vaccine With PO Cyclophosphamide | Total
Number analyzed (Participants) | 29 | 28 | 30 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 12 | 44
  >=65 years | 12 | 13 | 18 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.79 (10.83) | 64.96 (11.73) | 67.97 (9.96) | 65.28 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 16 | 37
  Male | 20 | 16 | 14 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 27 | 24 | 30 | 81
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 25 | 26 | 28 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Number of Participants With Treatment-related Grade 3 or 4 Local and Systemic Toxicity as Defined by NCI CTCAE v3.0
Time Frame: 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - GVAX Vaccine Without Cyclophosphamide | Arm B - GVAX Vaccine With IV Cyclophosphamide | Arm C - GVAX Vaccine With PO Cyclophosphamide
Number analyzed (Participants) | 29 | 28 | 30
Participants | 3 | 2 | 4

2. Primary Outcome: Amount of T-regulatory Cells (Tregs) and CD4+ and CD8+ Effector T Cells, After Neoadjuvant GVAX Pancreatic Cancer Vaccination.
Time Frame: up to 8 years
Population: Data was not collected for this outcome measure.
Arm/Group | Arm A - GVAX Vaccine Without Cyclophosphamide | Arm B - GVAX Vaccine With IV Cyclophosphamide | Arm C - GVAX Vaccine With PO Cyclophosphamide
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Change in the Number and Function of Peripheral Mesothelin-specific CD8+ T Cells and CD4+, FoxP3+, and GITR+ Tregs
Description: Change in the number and function of peripheral mesothelin-specific CD8+ T cells and CD4+, FoxP3+, and GITR+ Tregs after each GVAX pancreatic cancer vaccination when administered alone or in combination with a single dose or metronomic doses of cyclophosphamide.
Time Frame: up to 8 years
Population: Data was not collected for this outcome measure.
Arm/Group | Arm A - GVAX Vaccine Without Cyclophosphamide | Arm B - GVAX Vaccine With IV Cyclophosphamide | Arm C - GVAX Vaccine With PO Cyclophosphamide
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Overall Survival
Description: OS will be measured from date of randomization until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 10 years and 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 29 | 28 | 30
months | 34.2 [21.6 to 45.7] | 15.4 [13.2 to 26.5] | 16.5 [11.3 to 25.2]

5. Secondary Outcome: Disease Free Survival
Description: Disease free survival is defined as the time interval from the date of randomization to the date of radiographic evidence of disease recurrence. Estimation based on the Kaplan-Meier curve.
Time Frame: 10 years and 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - GVAX Vaccine Without Cyclophosphamide | Arm B - GVAX Vaccine With IV Cyclophosphamide | Arm C - GVAX Vaccine With PO Cyclophosphamide
Number analyzed (Participants) | 29 | 28 | 30
months | 18.92 [13.87 to 34.1] | 8.54 [2.66 to 17.1] | 5.56 [3.67 to 14.0]

ADVERSE EVENTS:
Time Frame: Up to 8 years
Description: Adverse events were collected through protocol defined mechanisms (i.e. regular investigator assessments and regular laboratory testing)
Groups:
- Arm C - GVAX Vaccine With PO Cyclophosphamide: Patients receive GVAX pancreatic cancer vaccine ID on day 1 of Cycle 1 and low-dose oral cyclophosphamide twice daily on days 1-7. Patients undergo pancreaticoduodenectomy on day 15. Approximately 6-10 weeks after surgery, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21 (Cycle 2). Beginning approximately 1 month after vaccination, patients receive standard adjuvant chemoradiotherapy comprising gemcitabine, fluorouracil or capecitabine, and radiotherapy over 26-28 weeks. Beginning approximately 4-8 weeks after the completion of chemoradiotherapy, patients receive the vaccine on day 1 and low-dose oral cyclophosphamide twice daily on days 1-7 and 15-21. Treatment with the vaccine and cyclophosphamide repeats every 28 days for 4 additional cycles.
  GVAX pancreatic cancer vaccine: Given intradermally
  cyclophosphamide: Given IV (Arm B), given orally (Arm C)
Arm/Group | Arm A - GVAX Vaccine Without Cyclophosphamide | Arm B - GVAX Vaccine With IV Cyclophosphamide | Arm C - GVAX Vaccine With PO Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/28 | 1/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 29/29 | 28/28 | 30/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - GVAX Vaccine Without Cyclophosphamide (N=29) | Arm B - GVAX Vaccine With IV Cyclophosphamide (N=28) | Arm C - GVAX Vaccine With PO Cyclophosphamide (N=30)
Nausea (Gastrointestinal disorders) | 0 | 9 | 7
Chills (General disorders) | 5 | 0 | 5 — and administration site conditions
Fatigue (General disorders) | 11 | 7 | 9 — and administration site conditions
Fever (General disorders) | 7 | 3 | 4 — and administration site conditions
Lymphocyte count decreased (Investigations) | 0 | 6 | 11
White blood cell count decreased (Investigations) | 2 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Blister, vaccine site (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Skin hyperpigmentation, vaccine site (Skin and subcutaneous tissue disorders) | 7 | 5 | 3
Erythema, vaccine site (Skin and subcutaneous tissue disorders) | 29 | 28 | 30
Induration, vaccine site (Skin and subcutaneous tissue disorders) | 29 | 26 | 30
Pruritus, vaccine site (Skin and subcutaneous tissue disorders) | 24 | 23 | 24
Tenderness, vaccine site (Skin and subcutaneous tissue disorders) | 23 | 18 | 19
Hives (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Vaccine site flare (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Warmth, vaccine site (Skin and subcutaneous tissue disorders) | 15 | 17 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes